CLINICAL TRIAL: NCT04973722
Title: A Randomized, Double-blind, Parallel-group Study in Chinese Healthy Male Subjects to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety and Immunogenicity of LY06006 Versus Prolia Following Single-dose Subcutaneous Injection
Brief Title: A Study to Evaluate LY06006 and Prolia in Healthy Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Luye Pharma Group Ltd. (Industry)
Collaborators: Shan Dong Boan Biotechnology Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LY06006/CT-CHN-103
Record Dates: First submitted 2021-04-20; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Healthy Adults
Keywords: Compare; Pharmacokinetics; Pharmacodynamics; Safety; Immunogenicity; LY06006; Prolia; Healthy Adults
MeSH Terms: interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LY06006 (Experimental): 60 mg/1 ml, once every 6 months administered subcutaneously
  Interventions: Drug: LY06006
- Prolia (Active Comparator): 60 mg/1 ml, once every 6 months administered subcutaneously
  Interventions: Drug: Prolia

INTERVENTIONS:
Drug: LY06006 — 60 mg/1 ml, once every 6 months administered subcutaneously
  Other Names: subcutaneous injection of 60 mg
  Arms: LY06006
Drug: Prolia — 60 mg/1 ml, once every 6 months administered subcutaneously
  Other Names: Denosumab
  Arms: Prolia

SUMMARY:
A randomized, double-blind, parallel-group study in Chinese healthy male subjects to evaluate the pharmacokinetics, pharmacodynamics, safety and immunogenicity of LY06006 versus Prolia following single-dose subcutaneous injection

DETAILED DESCRIPTION:
Study Design:

The study is a randomized, double-blind, parallel-group study in healthy adult male subjects to evaluate the pharmacokinetics, pharmacodynamics, safety and immunogenicity of LY06006 versus Prolia following single-dose subcutaneous injection.

A total of 168 healthy male subjects will be randomized 1:1 to receive a single subcutaneous (s.c.) injection of 60mg of either LY06006 ( LY06006 , 60 mg/1mL , Shandong Luye Pharmaceutical Co., Ltd.) or Prolia (60 mg / 1 mL , Amgen Inc.). During the entire study period, blood samples should be collected according to the Schedule of Assessments for pharmacokinetic, pharmacodynamic and immunogenicity analysis, and safety assessments should be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed the informed consent form;
2. Healthy males，ages ≥18 to ≤50 years;
3. Body weight ≥58 to ≤68 kg and Body mass index (BMI) >18 to <28 kg/m2, body mass index (BMI) = weight ( kg ) / height 2 (m 2);
4. Normal or clinically acceptable vital signs, physical exams, laboratory tests, 12- lead ECG, abdominal color Doppler ultrasound, chest radiograph, etc. screening;
5. No pregnancy plans and voluntarily take effective contraceptive measures from the screening date to the end of the study .

Exclusion Criteria:

1. Prior diagnosis of bone disease, or any condition that will affect bone metabolism such as, but not limit to: malignant tumors ( including myeloma ), hypoparathyroidism / hyperthyroidism, hypothyroidism / hyperthyroidism, acromegaly, Cushing ' s syndrome, hypopituitarism, severe chronic obstructive pulmonary disease, rheumatoid arthritis, osteomalacia;
2. Prior history or current evidence of osteomyelitis or osteonecrosis of the jaw (ONJ), or risk factors for ONJ such as invasive dental surgery or jaw surgery during the trial, or unhealed dental or oral surgery wounds;
3. Recent bone fracture within 6 months;
4. Active and unhealed infections of the respiratory system, digestive system, urinary system, reproductive system, or skin;
5. Serum calcium of < Lower Limit of Normal (LLN) or > Upper Limit of Normal (ULN);
6. Prior use of medications affecting bone turnover before screening and for the duration of study, including but not limited to: denosumab, bisphosphonates or fluoride within 12 months, contraceptives containing estrogen, tibolone, estrogen, selective estrogen receptor modulators, aromatase inhibitors, calcitonin, strontium salts, parathyroid hormone (or derivatives), vitamin D supplements ( >1000 IU/ day), anabolic steroids, systemic glucocorticoids, calcitriol or similar, diuretics, anticonvulsants within 6 months; inhaled or topical glucocorticoid drugs within 2 weeks;
7. Allergy to more than two drugs or food, or allergy to the ingredients of the investigational medicinal product (IMP);
8. Blood donation or massive blood loss ( ≥200 mL ) within 3 months before screening ;
9. Any vaccination within 6 months before screening or for the duration of study;
10. Prior use of any prescription drugs, over-the-counter drugs, any vitamin products or herbal medicines within 14 days before screening ;
11. Intense physical exercise within 2 weeks before screening or for the duration of the study, or any other conditions affecting drug absorption, distribution, metabolism, and excretion;
12. Upon enquiry, prior smoke more than 5 cigarettes per day within 3 months before the study;
13. Upon enquiry, a history of alcohol abuse ( drinking more than 14 units of alcohol per week within the first three months prior to screening : 1 unit = 350 mL of beer, 45 mL of liquor, or 150 mL of wine ), or positive alcohol test;
14. Positive urine screen for drug or a history of drug abuse or drug use in the past five years upon questioning ;
15. Other diseases with clinical significance (such as nervous system, mental system , cardiovascular system, urinary system, digestive system, respiratory system, metabolic endocrine system, blood system, skin disease, immune disease, tumor, etc.);
16. Any of the following tests positive: hepatitis B surface antigen ( HBsAg ), hepatitis C antibody ( HCV-AB ), human immunodeficiency virus antigen antibody ( HIVAg / Ab ) and treponema pallidum antibody;
17. Acute diseases or concomitant medications from screening to IMP administration;
18. Consumption of any alcohol-containing products within 48 hours before administration of the IMP ;
19. Prior participation in clinical trials for denosumab or denosumab biosimilar products; current participation in other clinical studies, or receiving or have received any investigational drug within 3 months (or less than 5-half lives of that medication, whichever time period is longer) before receiving study drug ;
20. History of fainting blood or needles;
21. In the opinion of the investigator, others to be excluded.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
AUC 0- ∞ | 168 days
  Area under the concentration-time curve from time zero to infinity
C max | 168 days
  Maximum observed concentration
s-CTX | 168 days
  Percent change in serum s-CTX from baseline.
AUEC0-t | 168 days
  The pharmacodynamic parameters
Emax | 168 days
  The pharmacodynamic parameters
TEmax | 168 days
  The pharmacodynamic parameters

SECONDARY OUTCOMES:
Vital signs：Temperature | 168 days
  Safety measures
Vital signs：pulse | 168 days
  Safety measures
Vital signs： blood pressure | 168 days
  Safety measures
Vital signs： respiration | 168 days
  Safety measures
Physical examination：general | 168 days
  Safety measures
Physical examination：head and neck region | 168 days
  Safety measures
Physical examination：lymph gland | 168 days
  Safety measures
Physical examination： oral cavity | 168 days
  Safety measures
Physical examination：chest | 168 days
  Safety measures
Physical examination：belly | 168 days
  Safety measures
Physical examination：Extremities and spine | 168 days
  Safety measures
Physical examination：nervous system | 168 days
  Safety measures
Laboratory tests：hematology | 168 days
  Safety measures
Laboratory tests：chemistry | 168 days
  Safety measures
Laboratory tests：urinalysis | 168 days
  Safety measures
Laboratory tests：parathyroid hormone | 168 days
  Safety measures
Laboratory tests：thyroid function | 168 days
  Safety measures
Laboratory tests：abdomen ultrasound | 168 days
  Safety measures
Laboratory tests：chest radiography | 168 days
  Safety measures
Laboratory tests：coagulation function | 168 days
  Safety measures
Electrocardiogram (12-Lead ECG) | 168 days
  Safety measures
Adverse events(AEs) | 168 days
  Safety measures
ADA | 168 days
  The incidence and antibody titer of ADA
Nab | 168 days
  The incidence of Nab.

CONTACTS AND LOCATIONS:
Overall Officials: Guoping Yang, doctor, Principal Investigator — The Third Xiangya Hospital of Central South University
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang S, Yang X, Huang J, Yang S, Wu Q, Chen H, Wu S, Dou C, Yang G, Xiang Y. Pharmacokinetics, pharmacodynamics, safety, and immunogenicity of a biosimilar of denosumab (LY06006): a randomized, double-blind, single-dose, parallel-controlled clinical study in healthy Chinese subjects. Expert Opin Investig Drugs. 2022 Oct;31(10):1133-1142. doi: 10.1080/13543784.2022.2120389. Epub 2022 Sep 7. PMID 36045484